CLINICAL TRIAL: NCT00503126
Title: Bivalirudin (Angiomax®) As A Procedural Anticoagulant In The Pediatric Population Undergoing Intravascular Procedures For Congenital Heart Disease
Brief Title: Bivalirudin as a Procedural Anticoagulant in Pediatrics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-07-01
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Cardiology
Keywords: pediatrics; bivalirudin
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bivalirudin — anticoagulation
  Other Names: Angiomax/Angiox

SUMMARY:
Pharmacokinetics and safety of weight based bivalirudin in children

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant females, with an age range of birth to 16 years of age.
* Expected to undergo a percutaneous intravascular procedure for the management of congenital heart disease.
* Written informed consent from a legal guardian/parent.
* Life expectancy of at least 15 days at study entry.
* Assent of the patient if older than 8 years, whenever possible.

Exclusion Criteria:

* History of intracerebral bleed (neonates confirmed by an ultrasound head scan prior to procedure), or cerebral arteriovenous malformation or any prior bleed with neurological deficit.
* Gastrointestinal or genitourinary bleeding within the last 2 weeks excluding normal menstrual cycles.
* Cerebrovascular accident within 6 months, or any cerebrovascular accident with a residual neurological deficit.
* Known congenital or acquired bleeding or clotting disorder.
* Patients undergoing renal dialysis.*
* Weight < 2.5 kg.
* Confirmed pregnancy at time of enrollment or breast feeding (females of child-bearing potential).
* Known allergy to bivalirudin or hirudin-derived drugs, or known sensitivity to any component of bivalirudin (Angiomax®).
* Any condition that in the investigator's opinion would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.
* Participation in another investigational therapeutic drug or therapeutic device trial within 30 days of starting study.
* Patients who have been receiving warfarin (Coumadin®) therapy and whose INR is > 1.5.
* Patients who cannot be discontinued from UFH at least 30 minutes prior to study drug bolus.
* Patients who have received a dose of LMWH within 8 hours prior to study drug bolus.
* Patients previously enrolled in the study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
PK/PD and safety | 30 days

REFERENCES:
- [Derived] Forbes TJ, Hijazi ZM, Young G, Ringewald JM, Aquino PM, Vincent RN, Qureshi AM, Rome JJ, Rhodes JF Jr, Jones TK, Moskowitz WB, Holzer RJ, Zamora R. Pediatric catheterization laboratory anticoagulation with bivalirudin. Catheter Cardiovasc Interv. 2011 Apr 1;77(5):671-9. doi: 10.1002/ccd.22817. Epub 2011 Jan 4. PMID 21433272